CLINICAL TRIAL: NCT02288715
Title: Relationship of Cerebral Perfusion Pressure Variability to Sepsis-associated Encephalopathy
Status: Completed | Type: Observational
Sponsor: Kang Yan (Other)
Responsible Party: Sponsor-Investigator, Kang Yan, Director of Intensive Care Unit, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: CPPV-KYan1205
Record Dates: First submitted 2014-10-27; First posted 2014-11-11 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Sepsis
Keywords: cerebral perfusion pressure; septic encephalopathy
MeSH Terms: conditions — Sepsis; Sepsis-Associated Encephalopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SAE: patient who develop encephalopathy in the progress of sepsis
  Interventions: Other: no interventions
- non-SAE: patient who do not develop encephalopathy in the progress of sepsis
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions

SUMMARY:
The purpose of the study is to evaluate whether variability of CPP (cerebral perfusion pressure) is related to sepsis-associated encephalopathy and outcomes of patients with sepsis.

DETAILED DESCRIPTION:
Encephalopathy is a common complication of sepsis, impaired cerebrovascular autoregulation (AR) in patients with sepsis is considered related to Sepsis-associated encephalopathy (SAE). As AR is important in stabilizing the cerebral perfusion pressure, whether greater variability of CPP is related to SAE and mortality or not remains unclear. We conduct this study to evaluate the relationship between them.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms of sepsis, severe sepsis and septic shock
* age over 18 years

Exclusion Criteria:

* preexisting Neurological diseases
* traumatic brain injury
* intracranial infectious disease
* severe hepatic or renal dysfunction
* ICU discharge Within 72 hours
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients admit to the general ICU of an academic teaching hospital
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
relationship between cerebral perfusion pressure variability and sepsis-associated encephalopathy | cerebral perfusion pressure is assessed up to 72 hours
  To estimate CPP noninvasively, we will monitor the middle cerebral artery flow velocity of patients with sepsis using transcranial Doppler ultrasound in the first 72h of their enrollment. Diagnosis of a SAE was performed using the confusion assessment method for ICU(CAM-ICU).

SECONDARY OUTCOMES:
Duration of mechanical ventilation | All the participants will be followed up until discharge or death, assessed up to 24 months
Time of ICU stay | All the participants will be followed up until discharge or death, assessed up to 24 months
Time of hospital stay | All the participants will be followed up until discharge or death, assessed up to 24 months
90-day mortality rate | All the participants will be followed up until 90 days after their enrollment or death
1-year mortality rate | All the participants will be followed up until 1 year after their enrollment or death
2-year mortality rate | All the participants will be followed up until 2 years after their enrollment or death
1-year quality of life of survivors | All the participants will be followed up until 1 year after their enrollment or death
  EQ-5D will be used to evaluate quality of life of survivors
2-year quality of life of survivors | All the participants will be followed up until 2 year after their enrollment or death
  EQ-5D will be used to evaluate quality of life of survivors

CONTACTS AND LOCATIONS:
Locations (1):
- Kang Yan, Chengdu, Sichuan, China